CLINICAL TRIAL: NCT05644808
Title: Molecularly Informed Lung Cancer Treatment in a Community Cancer Network: A Pragmatic Prospective RWE Study (MYLUNG Consortium: Part 2)
Brief Title: MYLUNG Consortium Study Protocol 2
Acronym: MYLUNG
Status: Active, not recruiting | Type: Observational
Sponsor: US Oncology Research (Industry)
Responsible Party: Sponsor
Other Study IDs: 20381
Record Dates: First submitted 2022-11-30; First posted 2022-12-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small Cell Lung Carcinoma; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer; Lung Cancer; Squamous Non-small Cell Lung Cancer; Non-squamous Non-small Cell Lung Cancer; Biomarker Testing; Tumor Tissue Testing
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-small Cell Lung Cancer

SUMMARY:
This pragmatic study looks to quantify the testing timeline, operational barriers, and outcomes of biomarker-guided therapy in a large, community-based, and largely unselected patient population with early stage and advanced stage, treatment-naive non-small cell lung cancer, whether squamous or non-squamous.

DETAILED DESCRIPTION:
Lung cancer remains the most lethal malignancy in men and women in the U.S. Providing high quality management of these patients in the community setting as compared to hospital or academic centers offers the opportunity to reduce cost without sacrificing clinical outcome and simultaneously improving patient convenience and value. Many patients diagnosed with late-stage cancers can benefit from advanced biomarker testing, yet not all eligible patients receive this type of diagnostic testing today.

Within advanced non-small-cell lung cancer (aNSCLC), there are many specific somatic mutations observed in select patient populations that have targeted highly effective and less toxic therapies. National guidelines have advocated for broad tumor molecular profiling as a part of the standard diagnostic evaluation for aNSCLC, with the goal of identifying driver mutations for which effective therapies or clinical trials are available.

Furthermore, there is emerging evidence that molecular testing can impact treatment choices in earlier stages of lung cancer. However, adherence to genomic testing guidelines presents unique challenges to community oncologists. While most oncology clinical research has been conducted at well-established academic medical centers, over 85% of cancer patients are diagnosed and treated at local, community-based clinical practices. Barriers exist in the ability to order these tests efficiently, in a timely manner, and reimbursed accordingly. Furthermore, patient care can vary drastically based on community-associated disparities.

This pragmatic clinical trial will generate Real World Evidence (RWE) to validate efficacy of first treatment regimen in newly diagnosed patients with non-small cell lung cancer. The MYLUNG Program integrates three separate protocols: Protocol #1 will interrogate historical data from a large number of practices seeing lung cancer patients to evaluate biomarker testing, decision making patterns, the patient journey, and the tissue journey; Protocol #2 (current trial) will prospectively evaluate the patient journey in a limited number of index practices focused on testing; integration of testing results; and treatments. Interventional strategies to optimize these objectives will be developed and integrated into Protocol #3, which will evaluate the impact of these strategies on the patient journey as it relates to shared decision making.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years and older) with newly diagnosed early stage, locally advanced or metastatic non-small cell lung cancer
* Eligible for systemic therapy based on the treating provider's assessment
* Subjects who developed locally advanced or metastatic disease after receiving adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the development of locally advanced or metastatic disease
* Subjects may be enrolled within 30 days of initiation of systemic therapy
* Signed informed consent

Exclusion Criteria:

* Stage IA at the time of enrollment
* Subjects with small cell lung cancer
* Subjects with Unknown primary tumor origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This pragmatic study looks to quantify the testing timeline, operational barriers, and outcomes of biomarker-guided therapy in a large, community-based, and largely unselected patient population with early stage and advanced stage, treatment naive non-small cell lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Who Do and Do Not Receive Biomarker Test Results Prior to Systemic Therapy or Death | 5 years from date of enrollment into study
  i. Comprehensive testing is defined as both PD-L1 testing to guide use of immunotherapies & testing for all genomic alterations for which we have FDA-approved therapies incl EGFR, ALK, ROS1, BRAF, NTRK, RET, KRAS & MET ii. Document whether patient receives single gene testing for actionable mutations compared to those who receive comprehensive testing. For patients who start systemic therapy prior to or without biomarker results, we will catalog reasons for not conducting testing incl:
  1. Clinical deterioration, clinical crisis
  2. Insufficient tissue
  3. Barriers to test ordering
     1. Tissue: obtaining sample, tissue retrieval
     2. Assay failure for 1 or more biomarkers: Quantity Not Sufficient (QNS), QA fail, test failure
     3. Patient/provider attitudes & perceptions
     4. Provider knowledge about testing options
     5. Patient knowledge about biomarker testing
     6. Payor Coverage: prior authorization denial, payor refusal
     7. Financial barriers: uncovered costs, reimbursement

SECONDARY OUTCOMES:
Proportion of patients placed on biomarker-directed first treatment regimen vs those who were not | 5 years from date of enrollment into study
  To determine the proportion of patients placed on biomarker-directed first treatment regimen. For patients who have received biomarker test results with at least one actionable mutation, catalog the reason for not prescribing biomarker-targeted therapy.
  i. Lack of availability or delays in obtaining targeted therapy ii. Misinterpretation of test results iii. Clinical contraindications (allergies, end organ dysfunction, active autoimmune disease, etc.) iv. Patient/provider attitudes and perceptions v. Financial barriers / Uncovered costs vi. Patient performance status
Time span between first systemic therapy as compared to date of initial presentation, date of diagnostic biopsy, date of first visit to a medical oncologist, and date of biomarker test order(s) and result(s). | 5 years from date of enrollment into study
Determine the variance in biomarker test order practice patterns by community cancer clinic settings as measured by percentage of comprehensive testing ordered, type of test ordered, and resulting treatment assigned to the patient. | 5 years from date of enrollment into study
  Characteristics of the cancer care practices include, but not limited to, number of geographic clinic locations, clinical settings (rural or urban), staffing and responsibilities, patient volumes, and Oncology Care Model (OCM) status.

CONTACTS AND LOCATIONS:
Overall Officials: Makenzi Evangelist, MD, Principal Investigator — New York Oncology Hematology
Locations (18):
- United States (18):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Illinois Cancer Specialists, Niles, Illinois
  - Maryland Oncology Hematology, P.A., Silver Spring, Maryland
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - New York Oncology Hematology, P.C., Albany, New York
  - Oncology Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Texas Oncology - West Texas, Abilene, Texas
  - Texas Oncology- DFWW, Arlington, Texas
  - Texas Oncology-Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-McAllen, McAllen, Texas
  - Texas Oncology- Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia